CLINICAL TRIAL: NCT07062952
Title: Kidney-protective Intervention With Salt Substitute After Kidney Tumor Surgery: a Single-center Randomized Controlled Study(KISS Study)
Brief Title: Kidney-protective Intervention With Salt Substitute After Kidney Tumor Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Le Qu, Associate chief urologist, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025DZKY-068-01
Record Dates: First submitted 2025-07-01; First posted 2025-07-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Kidney Tumors; CKD; Salt Substitute; Nephrectomy; eGFR
Keywords: kidney tumor; CKD; Salt substitute; nephrectomy; eGFR; kidney protection; kidney function; open-label; randomized controlled trial; Renal function compensation; CKD with clinical significance
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salt substitute (Experimental): Participants will consume salt substitutes
  Interventions: Dietary Supplement: Salt substitute
- Common salt (No Intervention): Participants will consume Common salt

INTERVENTIONS:
Dietary Supplement: Salt substitute — Patient consume salt substitutes daily while strictly adhering to WHO-recommendedsalt intake levels for 1 year.Salt substitutes (potassium-enriched low-sodium salt, primarily NaCl and KCl) reduce sodium content versus regular salt
  Arms: Salt substitute

SUMMARY:
This clinical trial is an open-label, randomized controlled study designed to evaluate the efficacyand safety of salt substitutes in protecting renal function after kidney tumor surgery, aiming toprovide dietary renal protection strategies for postoperative kidney tumor patients. lt will alsoassess the feasibility of salt substitute intervention. The primary research questions are:

1. Does a salt substitute diet significantly improve estimated glomerular filtration rate (eGFR) compared to a regular salt diet in postoperative kidney tumor patients?
2. What is the safety profile of salt substitute intervention in postoperative kidney tumor patients?
3. What is the compliance rate among postoperative kidney tumor patients using saltsubstitutes?
4. ls the salt substitute intervention feasible?

Researchers will compare the intervention group (salt substitute diet) with the control group (regular salt diet) to determine whether salt substitutes effectively improve postoperative eGFR in kidney tumor patients.

Participants will be required to:

1. Consume salt substitutes or regular salt daily while strictly adhering to WHO-recommendedsalt intake levels for 1 year.
2. Undergo scheduled baseline assessments at 1, 3, 6, and 12 months post-surgery, with 24-hoururine tests at months 1 and 6 to evaluate compliance.
3. Receive regular monitoring of blood electrolytes, eGFR, and other renal function indicators.
4. Document any adverse events or health status changes during the study period.

DETAILED DESCRIPTION:
Patients after kidney tumor surgery (radical nephrectomy or partial nephrectomy) experience acute loss of functional nephrons, causing compensatory hyperfunction in remaining nephrons under overload conditions. This manifests as elevated glomerular filtration rate (hyperfiltration), increased plasma flow (hyperperfusion), and heightened capillary transmembrane pressure (hypertension), collectively termed the "three-high glomerular state," significantly increasing risks of Acute Kidney Injury(AKI) and long-term Chronic Kidney Disease(CKD). Chinese populations consume salt far exceeding WHO recommendations, with proven associations to hypertension, stroke, cardiovascular disease, kidney disease, and gastric cancer. High salt intake elevates CKD risk through two pathways: chronic high salt consumption induces hypertension (a key CKD risk factor), and activates renal renin-angiotensin-aldosterone system (RAAS), promoting inflammation, fibrosis, and oxidative stress-induced kidney damage-exacerbating the postoperative "three-high state" and further increasing CKD risk. Additionally, Asian populations frequently carry salt-sensitive genetic variants, where both salt sensitivity and high intake cause mineralocorticoid receptor overactivation, independently amplifying CKD susceptibility. Salt substitutes (potassium-enriched low-sodium salt, primarily NaCl and KCl) reduce sodium content versus regular salt, potentially improving renal hemodynamics by lowering sodium load and supplementing potassium to delay renal function decline. Recent multicenter RCTs and meta-analyses confirm cardiovascular benefits: the SSaSS trial demonstrated 13% reduced cardiovascular event risk with potassium-enriched salt (25% KCl), preventing ~460,000 cardiovascular deaths annually via blood pressure control and ~743,000 non-fatal cardiovascular events (including ~120,000 CKD cases) without significant hyperkalemia-related adverse events. The DECIDESalt trial showed significant blood pressure reductions (SBP: -7.1 mmHg; DBP: -1.9 mmHg) and lower cardiovascular risk with salt substitutes versus regular salt, with post hoc analysis indicating reduced hypertension incidence in normotensive individuals without inducing hypotension. Meta-analyses highlight amplified benefits in high-risk populations and Asian diets via sodium-potassium homeostasis and vascular improvement, with clinically insignificant mild potassium elevation confirming efficacy and safety. Despite these cardiovascular benefits, salt substitutes' renal safety and efficacy in post-nephrectomy patients remain unreported. Thus, the investigators propose this open-label randomized controlled trial to evaluate salt substitutes for postoperative renal protection in kidney tumor patients, establishing evidence-based dietary strategies for renal function preservation.

Therefore, the investigators plan to provide study participants with free salt substitute and standardized salt containers (5g) for one year. Participants will receive a one-month supply of free salt substitute upon hospital discharge. Adherence will be assessed at the one-month follow-up visit via 24-hour urine collection. Based on adherence confirmation, the next two-month supply of free salt substitute will be dispensed, continuing until the three-month follow-up.

This process will be repeated for subsequent phases: Adherence will be evaluated at discharge and each follow-up visit before dispensing the next phase's supply of free salt substitute.To enhance adherence during the extended interval between the 6-month and 12-month postoperative follow-ups: A telemedicine follow-up will be conducted at 9 months post-operation.Adherence will be assessed using a self-administered questionnaire, and the salt substitute will be remotely dispensed upon confirmation.

Non-adherence protocol:

First occurrence: Participants will receive intensive education reinforcing the importance of salt substitute use to improve adherence.

Recurrence: Participants will be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following criteria:

  1. Voluntary participation with signed informed consent from both the primary participant and all cohabiting family members, with commitment to study procedures and follow-up;
  2. Age ≥18 years at enrollment (when signing informed consent), any gender;
  3. Diagnosed kidney tumor patients who underwent radical nephrectomy or partial nephrectomy (no restrictions on surgical approach);
  4. Preoperative eGFR >60 ml/min/1.73m² (calculated by CKD-EPI equation);
  5. Serum potassium <4.8 mmol/L;
  6. Predominantly home-based dietary habits (>90% meals prepared at home, assessed via self-report);
  7. Normal contralateral renal function at screening;
  8. Normal cardiopulmonary and hepatic function:

Exclusion Criteria:

* Participants will be excluded if they meet any of the following:

  1. Participant or cohabiting family members currently using potassium-sparing diuretics or potassium supplements, or prior use of salt substitutes;
  2. Post-discharge eGFR <45 ml/min/1.73m² without significant fluctuation;
  3. Comorbid chronic kidney diseases (e.g., diabetic nephropathy, lupus nephritis);
  4. Preoperative history of urinary tract obstruction;
  5. Cohabiting family member(s) with CKD (eGFR <45 ml/min/1.73m²);
  6. Planned postoperative nephrotoxic medications (e.g., anti-neoplastic agents, immunotherapy);
  7. Uncontrolled diabetes (HbA1c ≥12%);
  8. Uncontrolled hypertension (seated SBP ≥180 mmHg or DBP ≥110 mmHg), symptomatic hypotension (SBP <90 mmHg), or clinically evident hypovolemia;
  9. Preoperative proteinuria (≥1+ on dipstick);
  10. Severe cardiovascular disease (NYHA Class III-IV), gastrointestinal obstruction, or hyperkalemia history;
  11. BMI <18.5 kg/m² or >30 kg/m²;
  12. Participation in another clinical trial ≤30 days before randomization or concurrently;
  13. Communication barriers or anticipated non-adherence;
  14. Structural/functional urological abnormalities (e.g., duplicated kidneys, polycystic kidneys, renal artery stenosis, stones, BPH) or indwelling catheters;
  15. Prior radiotherapy/ablation/surgery on the contralateral kidney;
  16. Life expectancy <6 months (e.g., metastatic renal carcinoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) | Postoperative 12 months
  Estimated glomerular filtration rate (eGFR) in kidney tumor patients at 12 months after surgery

SECONDARY OUTCOMES:
Annual eGFR decline rate | Postoperative 12 months
  Annual decline rate of eGFR at 12 months postoperatively compared to the "new baseline" post-surgery
eGFR decline | Postoperative 12 months
  Proportion of patients with rapid eGFR decline (>3 ml/min/1.73m²/year) in each group
Reduction from baseline | Postoperative 12 months
  Decline in eGFR at 12 months postoperatively from the new postoperative baseline (ml/min/1.73m²)
Incidence of adverse events | Postoperative 12 months
  Incidence rate of hyperkalemia (serum potassium ≥5.5 mmol/L) and other adverse events
Incidence of CKD progression | Postoperative 12 months
  The 1-year incidence of CKD progression, which was defined as a worse CKD stage compared to baseline.
Progression of proteinuria | Postoperative 12 months
  Progression of proteinuria (defined as ≥30% increase in urine albumin-to-creatinine ratio from baseline)
Quality of life questionnaire score | Postoperative 12 months
  Kidney Disease Quality of Life 36-Item Short Form Survey;The scoring ranges from 0 to 100, with higher scores indicating better quality of life in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Nanjing, Jiangsu, China